CLINICAL TRIAL: NCT00846768
Title: Randomised, Double-Blind, Cross-over Study to Determine the 24-hour FEV1-time Profile of Orally Inhaled BI 1744 CL, Delivered With the Respimat Inhaler, After 3 Weeks of Once Daily or Twice Daily Administration in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: BI 1744 CL With Respimat Once Daily Versus Twice Daily in COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Crossover | Purpose: Treatment
Other Study IDs: 1222.26; EudtaCT No: 2008-006334-10
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol

INTERVENTIONS:
Drug: BI 1744 CL

SUMMARY:
The primary objective of the trial is to determine the effect of BI 17444Cl on the lung function over a 24-hour period, when it is inhaled using the Respimat inhaler in patients with chronic obstructive pulmonary disease. In the trial four treatments of each 3 weeks of duration are included: 2 dosages in a once daily administration and 2 dosages for administration twice daily.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent consistent with ICH-GCP guidelines prior to participation in the trial, which includes medication washout and restrictions
2. All patients must have a diagnosis of COPD and must meet the following spirometric criteria:

   Patients must have relatively stable airway obstruction with a post-bronchodilator FEV1 < 80% of predicted normal and a post-bronchodilator FEV1 / FVC < 70% at Visit 1
3. Male or female patients, 40 years of age or older
4. Patients must be current or ex-smokers with a smoking history of more than 10 pack years
5. Patients must be able to perform technically acceptable pulmonary function tests
6. Patients must be able to inhale medication in a competent manner from the Respimat inhaler and from a metered dose inhaler (MDI).

Exclusion Criteria:

1. Patients with a significant disease other than COPD.
2. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis; all patients with an SGOT > x2 ULN, SGPT > x2 ULN, bilirubin > x2 ULN or creatinine > x2 ULN will be excluded regardless of clinical condition.
3. Patients with a history of asthma. For patients with allergic rhinitis or atopy, source documentation is required to verify that the patient does not have asthma. If a patient has a total blood eosinophil count more than 600/mm3, source documentation is required to verify that the increased eosinophil count is related to a non-asthmatic condition.
4. Patients with any respiratory infection or COPD exacerbation in the 6 weeks prior to the Screening Visit (Visit 1) or during the baseline period.
5. Patients with any of the following conditions: a diagnosis of thyrotoxicosis; a diagnosis of paroxysmal tachycardia (>100 beats per minute)
6. Patients with any of the following conditions: a history of myocardial infarction within 1 year of screening visit (Visit 1); unstable or life-threatening cardiac arrhythmia; have been hospitalized for heart failure within the past year; known active tuberculosis; a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years (patients with treated basal cell carcinoma are allowed); a history of life-threatening pulmonary obstruction; a history of cystic fibrosis; clinically evident bronchiectasis; a history of significant alcohol or drug abuse
7. Patients who have undergone thoracotomy with pulmonary resection
8. Patients being treated with any of the following concomitant medications: oral beta2-adrenergics; oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
9. Patients who regularly use daytime oxygen therapy for more than one hour per day.
10. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the Screening Visit (Visit 1) or patients who are currently in a pulmonary rehabilitation program
11. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening Visit
12. Patients with known hypersensitivity to beta-adrenergics drugs, BAC, EDTA or any other component of the Respimat inhalation solution delivery system
13. Pregnant or nursing women
14. Women of childbearing potential not using two effective methods of birth control (one barrier, one non-barrier). Female patients will be considered to be of childbearing potential unless surgically sterilised by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years
15. Patients who have previously been randomized in this study or are currently participating in another study
16. Patients who are unable to comply with pulmonary medication restrictions prior to randomization

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- Belgium (3):
  - 1222.26.32008 Boehringer Ingelheim Investigational Site, Genk
  - 1222.26.32006 Boehringer Ingelheim Investigational Site, Ghent
  - 1222.26.32007 Boehringer Ingelheim Investigational Site, Hasselt
- Netherlands (2):
  - 1222.26.31002 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1222.26.31001 Boehringer Ingelheim Investigational Site, Heerlen

REFERENCES:
- [Derived] Joos GF, Aumann JL, Coeck C, Korducki L, Hamilton AL, Kunz C, Aalbers R. A randomised, double-blind, four-way, crossover trial comparing the 24-h FEV1 profile for once-daily versus twice-daily treatment with olodaterol, a novel long-acting beta2-agonist, in patients with chronic obstructive pulmonary disease. Respir Med. 2015 May;109(5):606-15. doi: 10.1016/j.rmed.2015.02.005. Epub 2015 Feb 14. PMID 25776199

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a multi-centre, randomised, double-blind, 4-way crossover trial. The duration of each treatment period was 3 weeks with no washout period between treatments.
Groups:
- Olo 2mcg Bid / Olo 10mcg qd / Olo 5mcg qd / Olo 5mcg Bid: Patients were administered Olodaterol 2 mcg bid in the first period, Olodaterol 10 mcg qd in the second period, Olodaterol 5 mcg qd in the third period and Olodaterol 5 mcg bid in the fourth period. Olodaterol was administered via the Respimat inhaler.
- Olo 5mcg qd / Olo 2mcg Bid / Olo 5mcg Bid / Olo 10mcg qd: Patients were administered Olodaterol 5 mcg qd in the first period, Olodaterol 2 mcg bid in the second period, Olodaterol 5 mcg bid in the third period and Olodaterol 10 mcg qd in the fourth period. Olodaterol was administered via the Respimat inhaler.
- Olo 5mcg Bid / Olo 5mcg qd / Olo 10mcg qd / Olo 2mcg Bid: Patients were administered Olodaterol 5 mcg bid in the first period, Olodaterol 5 mcg qd in the second period, Olodaterol 10 mcg qd in the third period and Olodaterol 2 mcg bid in the fourth period. Olodaterol was administered via the Respimat inhaler.
- Olo 10mcg qd / Olo 5mcg Bid / Olo 2mcg Bid / Olo 5mcg qd: Patients were administered Olodaterol 10 mcg qd in the first period, Olodaterol 5 mcg bid in the second period, Olodaterol 2 mcg bid in the third period and Olodaterol 5 mcg qd in the fourth period. Olodaterol was administered via the Respimat inhaler.
Period: Overall Study
Arm/Group | Olo 2mcg Bid / Olo 10mcg qd / Olo 5mcg qd / Olo 5mcg Bid | Olo 5mcg qd / Olo 2mcg Bid / Olo 5mcg Bid / Olo 10mcg qd | Olo 5mcg Bid / Olo 5mcg qd / Olo 10mcg qd / Olo 2mcg Bid | Olo 10mcg qd / Olo 5mcg Bid / Olo 2mcg Bid / Olo 5mcg qd
Started | 11 | 12 | 12 | 12
Completed | 11 | 11 | 12 | 12
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set, includes all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Study Total: Total number of patients treated in the study. This was a randomised, double-blind, active-controlled, 4 way crossover trial. 47 patients were assigned randomly to one of 4 treatment sequences in which they received each of the 4 treatments. The duration of each treatment period was 3 weeks with no washout period between treatments.
Arm/Group | Study Total
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.57 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: FEV1 Area Under Curve 0-12 h (AUC 0-12h) Response After 3 Weeks of Treatment
Description: Response was defined as change from baseline. Baseline FEV1 AUC (0-12) was defined as the AUC performed on the baseline visit, prior to the first dose of randomized treatment. FEV1 AUC 0-12h was calculated from 0-12 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: Day 0: -0:10, 0:30, 1, 2, 3, 4, 6, 8, 10, 11:50 h relative to planned morning dose on day 1; Day 21: -0:10, 0:30, 1, 2, 3, 4, 6, 8, 10, 11:50 h relative to morning dose
Population: Full analysis set (FAS). FAS is defined as all randomised and treated patients with baseline (pre-dose) data and evaluable post-dose data for at least one period.
Measure: Least Squares Mean (Standard Error); unit: Liter
Groups:
- Olo 2 mcg Bid: Olodaterol 2 mcg bid delivered by the Respimat Inhaler.
- Olo 5 mcg qd: Olodaterol 5 mcg qd delivered by the Respimat Inhaler.
- Olo 5 mcg Bid: Olodaterol 5 mcg bid delivered by the Respimat Inhaler.
- Olo 10 mcg qd: Olodaterol 10 mcg qd delivered by the Respimat Inhaler.
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 46 | 47 | 46 | 46
Liter | 0.155 (0.024) | 0.209 (0.024) | 0.189 (0.024) | 0.204 (0.024)
Statistical Analysis 1: Comparison: Olo 5 mcg Bid vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.3011, Mixed Models Analysis; Means adjusted using a mixed effects model with treatment and period as fixed effects and period as repeated effect with patient as repeated subject; Mean Difference (Final Values) = 0.015, 95% CI [-0.014 to 0.044], Standard Error of Mean 0.015 — Olo 10 mcg qd minus Olo 5 mcg bid
Statistical Analysis 2: Comparison: Olo 5 mcg qd vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.1582, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.021, 95% CI [-0.008 to 0.050], Standard Error of Mean 0.015 — Olo 5 mcg qd minus Olo 5 mcg bid
Statistical Analysis 3: Comparison: Olo 2 mcg Bid vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.054, 95% CI [0.025 to 0.083], Standard Error of Mean 0.015 — Olo 5 mcg qd minus Olo 2 mcg bid
Statistical Analysis 4: Comparison: Olo 5 mcg qd vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.7046, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.006, 95% CI [-0.034 to 0.023], Standard Error of Mean 0.015 — Olo 10 mcg qd minus Olo 5 mcg qd
Statistical Analysis 5: Comparison: Olo 2 mcg Bid vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.0248, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.033, 95% CI [0.004 to 0.063], Standard Error of Mean 0.015 — Olo 5 mcg bid minus Olo 2 mcg bid

2. Primary Outcome: FEV1 Area Under Curve 12-24 h (AUC 12-24h) Response After 3 Weeks of Treatment
Description: Response was defined as change from baseline. Baseline FEV1 AUC (12-24) was defined as the AUC performed on the baseline visit, prior to the first dose of randomized treatment. FEV1 AUC 12-24h was calculated from 12-24 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: Day 0: -0:10, 0:30, 1, 2, 10, 11, 11:50 h relative to planned evening dose on day 1; Day 21: -0:10, 0:30, 1, 2, 10, 11, 11:50 h relative to evening dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 46 | 47 | 46 | 46
Liter | 0.167 (0.022) | 0.155 (0.022) | 0.201 (0.022) | 0.149 (0.022)
Statistical Analysis 1: Comparison: Olo 5 mcg Bid vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.052, 95% CI [-0.081 to -0.023], Standard Error of Mean 0.015 — Olo 10 mcg qd minus Olo 5 mcg bid
Statistical Analysis 2: Comparison: Olo 5 mcg qd vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.047, 95% CI [-0.076 to -0.017], Standard Error of Mean 0.015 — Olo 5 mcg qd minus Olo 5 mcg bid
Statistical Analysis 3: Comparison: Olo 2 mcg Bid vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.4111, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.012, 95% CI [-0.041 to 0.017], Standard Error of Mean 0.015 — Olo 5 mcg qd minus Olo 2 mcg bid
Statistical Analysis 4: Comparison: Olo 5 mcg qd vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.7090, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.006, 95% CI [-0.035 to 0.024], Standard Error of Mean 0.015 — Olo 10 mcg qd minus Olo 5 mcg qd
Statistical Analysis 5: Comparison: Olo 2 mcg Bid vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.0211, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.035, 95% CI [0.005 to 0.064], Standard Error of Mean 0.015 — Olo 5 mcg bid minus Olo 2 mcg bid

3. Secondary Outcome: FEV1 Area Under Curve 0-24 h (AUC 0-24h) Response After 3 Weeks of Treatment
Description: Response was defined as change from baseline. Baseline FEV1 AUC (0-24) was defined as the AUC performed on the baseline visit, prior to the first dose of randomized treatment. FEV1 AUC 0-24h was calculated from 0-24 hours post-dose using the trapezoidal rule, divided by the observation time (24h) to report in litres.
Time Frame: Day0:-0:10,0:30,1,2,3,4,6,8,10,11:50h relative to planned morning dose on day1,0:30,1,2,10,11,11:50h relative to planned evening dose on day1; Day21:-0:10,0:30,1,2,3,4,6,8,10,11:50h relative to morning dose,0:30,1,2,10,11,11:50h relative to evening dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 46 | 47 | 46 | 46
Liter | 0.160 (0.022) | 0.182 (0.022) | 0.195 (0.022) | 0.176 (0.022)
Statistical Analysis 1: Comparison: Olo 5 mcg Bid vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1753, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.019, 95% CI [-0.045 to 0.008], Standard Error of Mean 0.014 — Olo 10 mcg qd minus Olo 5 mcg bid
Statistical Analysis 2: Comparison: Olo 5 mcg qd vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.3444, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.013, 95% CI [-0.040 to 0.014], Standard Error of Mean 0.014 — Olo 5 mcg qd minus Olo 5 mcg bid
Statistical Analysis 3: Comparison: Olo 2 mcg Bid vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1161, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.022, 95% CI [-0.005 to 0.049], Standard Error of Mean 0.014 — Olo 5 mcg qd minus Olo 2 mcg bid
Statistical Analysis 4: Comparison: Olo 5 mcg qd vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.6789, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.006, 95% CI [-0.033 to 0.021], Standard Error of Mean 0.014 — Olo 10 mcg qd minus Olo 5 mcg qd
Statistical Analysis 5: Comparison: Olo 2 mcg Bid vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.0129, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.035, 95% CI [0.007 to 0.062], Standard Error of Mean 0.014 — Olo 5 mcg bid minus Olo 2 mcg bid

4. Secondary Outcome: Peak FEV1 (0-3h) Response After 3 Weeks
Description: Response was defined as change from baseline. Study baseline peak FEV1 was defined as the mean of the available pre-dose peak FEV1 values prior to first dose of treatment. Peak FEV1 (0-3h) values were obtained within 0 - 3 hours after the last dose after three weeks of treatment.
Time Frame: Baseline, 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 45 | 47 | 46 | 46
Liter | 0.187 (0.029) | 0.249 (0.029) | 0.230 (0.029) | 0.242 (0.029)
Statistical Analysis 1: Comparison: Olo 5 mcg Bid vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.4931, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.012, 95% CI [-0.023 to 0.047], Standard Error of Mean 0.017 — Olo 10 mcg qd minus Olo 5 mcg bid
Statistical Analysis 2: Comparison: Olo 5 mcg qd vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.2597, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.020, 95% CI [-0.015 to 0.054], Standard Error of Mean 0.017 — Olo 5 mcg qd minus Olo 5 mcg bid
Statistical Analysis 3: Comparison: Olo 2 mcg Bid vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.062, 95% CI [0.027 to 0.097], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Olo 2 mcg bid
Statistical Analysis 4: Comparison: Olo 5 mcg qd vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.6578, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.008, 95% CI [-0.042 to 0.027], Standard Error of Mean 0.017 — Olo 10 mcg qd minus Olo 5 mcg qd
Statistical Analysis 5: Comparison: Olo 2 mcg Bid vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.0175, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.042, 95% CI [0.008 to 0.077], Standard Error of Mean 0.018 — Olo 5 mcg bid minus Olo 2 mcg bid

5. Secondary Outcome: Trough FEV1 Response
Description: Response was defined as change from baseline. Study baseline trough FEV1 was defined as the mean of the available pre-dose trough FEV1 values prior to first dose of treatment. Trough values were the mean of values obtained 23h and 23 h 50 min after the last dose of study drug after three weeks of treatment .
Time Frame: Baseline, 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 45 | 47 | 46 | 46
Liter | 0.093 (0.028) | 0.108 (0.028) | 0.129 (0.028) | 0.087 (0.028)
Statistical Analysis 1: Comparison: Olo 5 mcg Bid vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0353, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.042, 95% CI [-0.081 to -0.003], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Olo 5 mcg bid
Statistical Analysis 2: Comparison: Olo 5 mcg qd vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.2875, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.021, 95% CI [-0.060 to 0.018], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Olo 5 mcg bid
Statistical Analysis 3: Comparison: Olo 2 mcg Bid vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.4553, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.015, 95% CI [-0.024 to 0.054], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Olo 2 mcg bid
Statistical Analysis 4: Comparison: Olo 5 mcg qd vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.2902, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.021, 95% CI [-0.060 to 0.018], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Olo 5 mcg qd
Statistical Analysis 5: Comparison: Olo 2 mcg Bid vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.0731, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.036, 95% CI [-0.003 to 0.075], Standard Error of Mean 0.020 — Olo 5 mcg bid minus Olo 2 mcg bid

6. Secondary Outcome: FVC Area Under Curve 0-12 h (AUC 0-12h) Response After 3 Weeks of Treatment
Description: Response was defined as change from baseline. Baseline FVC AUC (0-12) was defined as the AUC performed on the baseline visit, prior to the first dose of randomized treatment. FVC AUC 0-12h was calculated from 0-12 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 46 | 47 | 46 | 46
Liter | 0.262 (0.043) | 0.335 (0.043) | 0.294 (0.043) | 0.340 (0.043)
Statistical Analysis 1: Comparison: Olo 5 mcg Bid vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0917, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.046, 95% CI [-0.008 to 0.099], Standard Error of Mean 0.027 — Olo 10 mcg qd minus Olo 5 mcg bid
Statistical Analysis 2: Comparison: Olo 5 mcg qd vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.1273, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.041, 95% CI [-0.012 to 0.095], Standard Error of Mean 0.027 — Olo 5 mcg qd minus Olo 5 mcg bid
Statistical Analysis 3: Comparison: Olo 2 mcg Bid vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0080, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.073, 95% CI [0.019 to 0.127], Standard Error of Mean 0.027 — Olo 5 mcg qd minus Olo 2 mcg bid
Statistical Analysis 4: Comparison: Olo 5 mcg qd vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.8683, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.004, 95% CI [-0.049 to 0.058], Standard Error of Mean 0.027 — Olo 10 mcg qd minus Olo 5 mcg qd
Statistical Analysis 5: Comparison: Olo 2 mcg Bid vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.2444, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.032, 95% CI [-0.022 to 0.086], Standard Error of Mean 0.027 — Olo 5 mcg bid minus Olo 2 mcg bid

7. Secondary Outcome: FVC Area Under Curve 12-24 h (AUC 12-24h) Response After 3 Weeks of Treatment
Description: Response was defined as change from baseline. Baseline FVC AUC (12-24) was defined as the AUC performed on the baseline visit, prior to the first dose of randomized treatment. FVC AUC 12-24h was calculated from 12-24 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 46 | 47 | 46 | 46
Liter | 0.239 (0.043) | 0.215 (0.043) | 0.318 (0.043) | 0.219 (0.043)
Statistical Analysis 1: Comparison: Olo 5 mcg Bid vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0023, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.099, 95% CI [-0.162 to -0.036], Standard Error of Mean 0.032 — Olo 10 mcg qd minus Olo 5 mcg bid
Statistical Analysis 2: Comparison: Olo 5 mcg qd vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.103, 95% CI [-0.165 to -0.040], Standard Error of Mean 0.032 — Olo 5 mcg qd minus Olo 5 mcg bid
Statistical Analysis 3: Comparison: Olo 2 mcg Bid vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.4508, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.024, 95% CI [-0.087 to 0.039], Standard Error of Mean 0.032 — Olo 5 mcg qd minus Olo 2 mcg bid
Statistical Analysis 4: Comparison: Olo 5 mcg qd vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.9087, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.004, 95% CI [-0.059 to 0.066], Standard Error of Mean 0.032 — Olo 10 mcg qd minus Olo 5 mcg qd
Statistical Analysis 5: Comparison: Olo 2 mcg Bid vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.0146, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.079, 95% CI [0.016 to 0.142], Standard Error of Mean 0.032 — Olo 5 mcg bid minus Olo 2 mcg bid

8. Secondary Outcome: FVC Area Under Curve 0-24 h (AUC 0-24h) Response After 3 Weeks of Treatment
Description: Response was defined as change from baseline. Baseline FVC AUC (0-24) was defined as the AUC performed on the baseline visit, prior to the first dose of randomized treatment. FVC AUC 0-24h was calculated from 0-24 hours post-dose using the trapezoidal rule, divided by the observation time (24h) to report in litres.
Time Frame: Day0:-0:10,0:30,1,2,3,4,6,8,10,11:50h relative to planned morning dose on day1, 0:30,1,2,10,11,11:50h relative to planned evening dose on day1; Day21:-0:10,0:30,1,2,3,4,6,8,10,11:50h relative to morning dose,0:30,1,2,10,11,11:50h relative to evening dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 46 | 47 | 46 | 46
Liter | 0.249 (0.041) | 0.275 (0.041) | 0.306 (0.041) | 0.279 (0.041)
Statistical Analysis 1: Comparison: Olo 5 mcg Bid vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.3291, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.027, 95% CI [-0.080 to 0.027], Standard Error of Mean 0.027 — Olo 10 mcg qd minus Olo 5 mcg bid
Statistical Analysis 2: Comparison: Olo 5 mcg qd vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.2638, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.030, 95% CI [-0.084 to 0.023], Standard Error of Mean 0.027 — Olo 5 mcg qd minus Olo 5 mcg bid
Statistical Analysis 3: Comparison: Olo 2 mcg Bid vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.3386, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.026, 95% CI [-0.028 to 0.080], Standard Error of Mean 0.027 — Olo 5 mcg qd minus Olo 2 mcg bid
Statistical Analysis 4: Comparison: Olo 5 mcg qd vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.8877, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.004, 95% CI [-0.050 to 0.057], Standard Error of Mean 0.027 — Olo 10 mcg qd minus Olo 5 mcg qd
Statistical Analysis 5: Comparison: Olo 2 mcg Bid vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.0402, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.057, 95% CI [0.003 to 0.111], Standard Error of Mean 0.027 — Olo 5 mcg bid minus Olo 2 mcg bid

9. Secondary Outcome: Peak FVC (0-3h) Response After 3 Weeks
Description: Response was defined as change from baseline. Study baseline peak FVC was defined as the mean of the available pre-dose peak FVC values prior to first dose of treatment. Peak FVC (0-3h) values were obtained within 0 - 3 hours after the last dose after three weeks of treatment.
Time Frame: Baseline, 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 45 | 47 | 46 | 46
Liter | 0.325 (0.049) | 0.417 (0.049) | 0.349 (0.049) | 0.433 (0.049)
Statistical Analysis 1: Comparison: Olo 5 mcg Bid vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0133, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.084, 95% CI [0.018 to 0.151], Standard Error of Mean 0.034 — Olo 10 mcg qd minus Olo 5 mcg bid
Statistical Analysis 2: Comparison: Olo 5 mcg qd vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.0450, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.068, 95% CI [0.002 to 0.135], Standard Error of Mean 0.034 — Olo 5 mcg qd minus Olo 5 mcg bid
Statistical Analysis 3: Comparison: Olo 2 mcg Bid vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0078, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.092, 95% CI [0.025 to 0.159], Standard Error of Mean 0.034 — Olo 5 mcg qd minus Olo 2 mcg bid
Statistical Analysis 4: Comparison: Olo 5 mcg qd vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.6268, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.016, 95% CI [-0.050 to 0.083], Standard Error of Mean 0.034 — Olo 10 mcg qd minus Olo 5 mcg qd
Statistical Analysis 5: Comparison: Olo 2 mcg Bid vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.4891, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.024, 95% CI [-0.044 to 0.091], Standard Error of Mean 0.034 — Olo 5 mcg bid minus Olo 2 mcg bid

10. Secondary Outcome: Trough FVC Response
Description: Response was defined as change from baseline. Study baseline trough FVC was defined as the mean of the available pre-dose trough FVC values prior to first dose of treatment. Trough values were the mean of values obtained 23h and 23 h 50 min after the last dose of study drug after three weeks of treatment .
Time Frame: Baseline, 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 45 | 47 | 46 | 46
Liter | 0.111 (0.054) | 0.177 (0.054) | 0.181 (0.054) | 0.162 (0.054)
Statistical Analysis 1: Comparison: Olo 5 mcg Bid vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.6259, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.019, 95% CI [-0.097 to 0.059], Standard Error of Mean 0.040 — Olo 10 mcg qd minus Olo 5 mcg bid
Statistical Analysis 2: Comparison: Olo 5 mcg qd vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.9190, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.004, 95% CI [-0.082 to 0.074], Standard Error of Mean 0.039 — Olo 5 mcg qd minus Olo 5 mcg bid
Statistical Analysis 3: Comparison: Olo 2 mcg Bid vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0985, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.066, 95% CI [-0.012 to 0.145], Standard Error of Mean 0.040 — Olo 5 mcg qd minus Olo 2 mcg bid
Statistical Analysis 4: Comparison: Olo 5 mcg qd vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.6991, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.015, 95% CI [-0.093 to 0.063], Standard Error of Mean 0.039 — Olo 10 mcg qd minus Olo 5 mcg qd
Statistical Analysis 5: Comparison: Olo 2 mcg Bid vs Olo 5 mcg Bid; Test type: Superiority or Other; p = 0.0802, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.070, 95% CI [-0.009 to 0.149], Standard Error of Mean 0.040 — Olo 5 mcg bid minus Olo 2 mcg bid

11. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis, ECG and Physical Examination
Description: Clinical relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG. New abnormal findings or worsenings of baseline conditions were reported as Adverse Events related to treatment (cardiac disorders and investigations).
Time Frame: 3 weeks
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 47 | 47 | 46 | 46
percentage of participants
  Cardiac disorders | 0.0 | 0.0 | 0.0 | 0.0
  Investigations | 0.0 | 0.0 | 0.0 | 0.0

12. Secondary Outcome: Pharmacokinetics (PK): Concentration of the Analyte in Plasma Measured at 0.167 Hours Post Dosing at Steady State
Description: Steady state concentration of the analyte in plasma measured at 0.167 hours post dosing in week 3. The start of inhalation was used as time point 0 for calculation of pharmacokinetic parameters. Descriptive statistics were calculated only if N>=16 had concentrations within the validated concentration range.
Time Frame: 3 weeks
Population: All evaluable subjects. A subject was considered to be not evaluable if the subject had a protocol violation relevant to the evaluation of PK parameters or had insufficient data. In the "Olo 2 mcg Bid" Arm, there were only 14 patients with values within the validated concentration range.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 0 | 25 | 36 | 41
pg/mL |  | 3.52 (35.9) | 4.28 (42.0) | 5.78 (62.1)

13. Secondary Outcome: Pharmacokinetics (PK): Amount of Analyte That is Eliminated in Urine at Steady State From the Time Point 0 Hours to Time Point 12 Hours
Description: Amount of analyte that is eliminated in urine at steady state from the time point 0 hours to time point 12 hours after dosing in week 3 (after the morning dose for the bid dose regimens). The start of inhalation was used as time point 0 for calculation of pharmacokinetic parameters.
  Descriptive statistics were calculated only if N>=16 had concentrations within the validated concentration range.
Time Frame: 3 weeks
Population: All evaluable subjects. A subject was considered to be not evaluable if the subject had a protocol violation relevant to the evaluation of PK parameters or had insufficient data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 45 | 47 | 46 | 46
ng | 68.2 (67.5) | 115 (68.8) | 177 (64.8) | 213 (70.6)

14. Secondary Outcome: Pharmacokinetics (PK): Amount of Analyte That is Eliminated in Urine at Steady State From the Time Point 0 Hours to Time Point 24 Hours
Description: Amount of analyte that is eliminated in urine at steady state from the time point 0 hours to time point 24 hours after dosing in week 3. The start of inhalation was used as time point 0 for calculation of pharmacokinetic parameters. Descriptive statistics were calculated only if N>=16 had concentrations within the validated concentration range.
Time Frame: 3 weeks
Population: All evaluable subjects. A subject was considered to be not evaluable if the subject had a protocol violation relevant to the evaluation of PK parameters or had insufficient data.
  This endpoint was only calculated for the two qd dose regimens, therefore the number of patients in the Olo 2 Mcg Bid Arm and the Olo 5 Mcg Bid Arm is 0.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 0 | 46 | 0 | 46
ng |  | 181 (66.8) |  | 343 (65.9)

15. Secondary Outcome: Pharmacokinetics (PK): Fraction of Analyte Eliminated in Urine at Steady State From Time Point 0 Hours to Time Point 12 Hours
Description: Fraction of analyte eliminated in urine at steady state from time point 0 hours to time point 12 hours after dosing in week 3 (after the morning dose for the bid dose regimens). The start of inhalation was used as time point 0 for calculation of pharmacokinetic parameters.
  Descriptive statistics were calculated only if N>=16 had concentrations within the validated concentration range.
Time Frame: 3 weeks
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 45 | 47 | 46 | 46
percent | 3.41 (67.5) | 2.29 (68.8) | 3.55 (64.8) | 2.13 (70.6)

16. Secondary Outcome: Pharmacokinetics (PK): Fraction of Analyte Eliminated in Urine at Steady State From Time Point 0 Hours to Time Point 24 Hours
Description: Fraction of analyte eliminated in urine at steady state from time point 0 hours to time point 24 hours after dosing in week 3. The start of inhalation was used as time point 0 for calculation of pharmacokinetic parameters. Descriptive statistics were calculated only if N>=16 had concentrations within the validated concentration range.
Time Frame: 3 weeks
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 0 | 46 | 0 | 46
percent |  | 3.61 (66.8) |  | 3.43 (65.9)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Olo 2 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Serious Adverse Events (participants affected / at risk) | 1/47 | 0/47 | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 1/47 | 4/47 | 4/46 | 3/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olo 2 mcg Bid (N=47) | Olo 5 mcg qd (N=47) | Olo 5 mcg Bid (N=46) | Olo 10 mcg qd (N=46)
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olo 2 mcg Bid (N=47) | Olo 5 mcg qd (N=47) | Olo 5 mcg Bid (N=46) | Olo 10 mcg qd (N=46)
Nasopharyngitis (Infections and infestations) | 1 | 1 | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.